CLINICAL TRIAL: NCT04066348
Title: Clinical Trial of Etanercept (TNF-α Blocker) for Treatment of Blast-Induced Tinnitus
Brief Title: TNF-α Treatment of Blast-Induced Tinnitus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: University of Miami (Other); Michigan Ear Institute (Unknown)
Responsible Party: Principal Investigator, Dr. Jinsheng Zhang, Principle Investigator, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR172190
Record Dates: First submitted 2019-07-29; First posted 2019-08-26 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-05

CONDITIONS: Tinnitus, Noise Induced
Keywords: tinnitus; etanercept; tinnitus function index; tinnitus primary function; audiological evaluation
MeSH Terms: conditions — Tinnitus | interventions — Etanercept; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Etanercept Injection Group (Experimental): Subjects will receive 2 X 25mg/ 1ml etanercept injection (experimental) weekly for 12 weeks.
  Interventions: Biological: Etanercept
- Placebo Injection Group (Placebo Comparator): Subjects will receive 2 X 1ml saline injection (placebo) weekly for 12 weeks.
  Interventions: Other: Saline

INTERVENTIONS:
Biological: Etanercept — To treat blast or noise induced tinnitus
  Other Names: Enbrel
  Arms: Etanercept Injection Group
Other: Saline — Placebo
  Arms: Placebo Injection Group

SUMMARY:
The purpose of this multi-site research study is to determine if Etanercept, compared to a placebo, significantly reduces the severity of tinnitus (ringing in the ears) associated with history of blast and/or noise exposure or associated with Traumatic Brain Injury (TBI) and/or concussion. Individuals who qualify will be randomized into one of two groups: The group receiving the medication Etanercept or the group receiving a saline solution placebo.

DETAILED DESCRIPTION:
The primary objectives are to test if: 1) Etanercept significantly reduces tinnitus distress as measured by Tinnitus Functional Index (TFI); and 2) Etanercept improves hearing. In addition, the investigators will explore whether Etanercept treatment leads to sustained therapeutic effects over time;

The secondary objective is to test if: 1) Etanercept reduces tinnitus loudness measured by visual numeric scale (VNS) rating.

ELIGIBILITY:
Inclusion Criteria:

1. Tinnitus of at least a moderate severity as defined by a score of ≥ 25 points or higher on the Tinnitus Functional Index (TFI) questionnaire associated with one or more of the following:

   1. Blast- or noise exposure
   2. Traumatic brain injury (TBI) and/or concussion diagnosed by a health care provider.
2. Able to provide written informed consent.
3. Age: Minimum 18 years of age at the time of enrollment.
4. Other concurrent treatments for tinnitus: A four-week washout from any other tinnitus treatment or management program is required prior to entering this study.

   a) Hearing aids are permitted if the participant has been wearing them for at least 4 weeks.
5. Hearing function: All degrees of hearing function can be included, recognizing that individuals with profound, bilateral hearing loss will not be able to perform tinnitus evaluations and hearing tests but will be able to rate subjective tinnitus loudness, annoyance and impact on life. This is an important sub-population because of the challenges in treating them with acoustic therapy and the need for a medical intervention.
6. Additional tinnitus characteristics:

   a) Tinnitus history: Onset associated with blast and/or noise exposure or associated with diagnosed TBI and/or concussion. Subjects will have blast exposure, noise exposure, traumatic brain injury (TBI), and/or concussion impact, defined as exposure/impact less than or longer than six months at time of enrollment.

   i. Participants enrolled with tinnitus associated with TBI and/or concussion must have received a diagnosis of TBI and/or concussion by a health care provider.

   b) Stability: Constant (not pulsatile or intermittent). c) Location of tinnitus perception: Unrestricted. Tinnitus may be unilateral, bilateral, or perceived in the head.

Exclusion Criteria:

1. History or evidence of any of the following: Significant brain malformation; cerebral vascular events (such as strokes); neurodegenerative disorders affecting the brain, such as Parkinson's disease, ALS, or Huntington's disease; multiple sclerosis, Guillain-Barré syndrome, or any other disease involving demyelination disorder or any finding suggesting a demyelination disease or disorder; prior brain surgery.

   a. The following surgical procedures are not exclusionary: Evacuation of subdural hematoma, insertion of intracranial pressure monitor device, craniectomy
2. Active malignant neoplasm such as lymphoma or solid tumors or history of malignant neoplasm, excluding successfully treated squamous cell carcinoma or basal carcinoma of the skin or cervical cancer.
3. Diagnosis of congestive heart failure.
4. History of diagnosed seizure disorder or epilepsy.
5. Diagnosis of myelodysplastic syndrome or aplastic anemia, white blood cell count < 4000, or platelet count < 150,000.
6. Subjects who currently have an active infection, including tuberculosis, HIV, hepatitis B, and/or chicken pox.

   a. Patients with latent hepatitis B infection are also excluded from participation.
7. Scheduled to receive a live vaccine during study participation or received a live vaccine within 2 weeks prior to screening visit/procedures.
8. Diagnosis of an auto-immune disease that, in the opinion of the investigator, would cause a weakened immune system.

   a) Autoimmune thyroid disease is not considered an exclusionary autoimmune disease for participation in this study.
9. Diabetes.
10. Ongoing treatment with or plans to begin taking any of the following contraindicated medications: Cyclophosphamide or sulfasalazine; abatacept, anakinra, or any other immunomodulatory biologic therapy; sulfonylureas, meglitinides, or insulin.
11. Subjects who cannot communicate reliably with research team members or who are not likely to be able to complete the requirements of the trial per the discretion of the investigator.
12. Subjects who have participated in a drug clinical trial within the last 30 days before the start of this one.
13. Pregnancy or planned pregnancy during the study.
14. Women who are lactating or are of child-bearing-age without use of contraception.
15. MMSE score < 24.
16. Clinically significant out of range laboratory values for protocol required laboratory tests as assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Functional Index (TFI) | 12 Weeks
  Self-report questionnaire used to assess the severity and negative impact of tinnitus (tinnitus distress). It uses an 11 point Likert scale with higher scores indicating more severe tinnitus (For example, "How strong or loud was your tinnitus?", 0 (Not at all strong or loud)-10 (Extremely strong or loud).

SECONDARY OUTCOMES:
Audiometric testing | 12 Weeks
  Pure tone air conduction (AC) testing; Pure tone bone conduction (BC) testing; Speech recognition threshold (SRT); Tympanometry; Word recognition testing
Tinnitus Testing | 12 Weeks
  Tinnitus loudness matching (1 kHz loudness-matching); Minimum Masking Levels (MMLs)
Visual Numeric Rating Scale | 12 Weeks
  Self-rated visual numeric scale that asks respondents to rate the loudness of their tinnitus on a scale from 0 (No Tinnitus) to 10 (Very Loud). Higher scores indicate louder/more severe tinnitus.
Tinnitus Primary Function Questionnaire | 12 Weeks
  Self-report questionnaire assessing primary activities impaired by tinnitus. The questionnaire uses a self report number scale (1-100) asking respondents to indicate their agreement with each statement on a scale from 0 (completely disagree) to 100 (completely agree). Higher scores indicate worse tinnitus/more functional impairment from tinnitus.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsheng Zhang, Ph. D., Principal Investigator — Wayne State University
Locations (4):
- United States (4):
  - Advent Health, Celebration, Florida
  - University of Miami, Coral Gables, Florida
  - Wayne State University, Detroit, Michigan
  - Michigan Ear Institute, Farmington Hills, Michigan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Meikle MB, Henry JA, Griest SE, Stewart BJ, Abrams HB, McArdle R, Myers PJ, Newman CW, Sandridge S, Turk DC, Folmer RL, Frederick EJ, House JW, Jacobson GP, Kinney SE, Martin WH, Nagler SM, Reich GE, Searchfield G, Sweetow R, Vernon JA. The tinnitus functional index: development of a new clinical measure for chronic, intrusive tinnitus. Ear Hear. 2012 Mar-Apr;33(2):153-76. doi: 10.1097/AUD.0b013e31822f67c0. PMID 22156949
- [Background] Lew HL, Jerger JF, Guillory SB, Henry JA. Auditory dysfunction in traumatic brain injury. J Rehabil Res Dev. 2007;44(7):921-8. doi: 10.1682/jrrd.2007.09.0140. PMID 18075949
- [Background] VBA. VA Annual Benefits Report: Fiscal Year 2012. In: VA US, ed. 810 Vermont Avenue N. W. , Washington, D.C., 20420: Veterans Benefits Administration, 2013:82.
- [Background] Hesser H, Westin V, Hayes SC, Andersson G. Clients' in-session acceptance and cognitive defusion behaviors in acceptance-based treatment of tinnitus distress. Behav Res Ther. 2009 Jun;47(6):523-8. doi: 10.1016/j.brat.2009.02.002. Epub 2009 Feb 10. PMID 19268281
- [Background] Crocetti A, Forti S, Ambrosetti U, Bo LD. Questionnaires to evaluate anxiety and depressive levels in tinnitus patients. Otolaryngol Head Neck Surg. 2009 Mar;140(3):403-5. doi: 10.1016/j.otohns.2008.11.036. PMID 19248952
- [Background] Hasson D, Theorell T, Wallen MB, Leineweber C, Canlon B. Stress and prevalence of hearing problems in the Swedish working population. BMC Public Health. 2011 Feb 23;11:130. doi: 10.1186/1471-2458-11-130. PMID 21345187
- [Background] Hebert S, Fullum S, Carrier J. Polysomnographic and quantitative electroencephalographic correlates of subjective sleep complaints in chronic tinnitus. J Sleep Res. 2011 Mar;20(1 Pt 1):38-44. doi: 10.1111/j.1365-2869.2010.00860.x. PMID 20561177
- [Background] Stevens C, Walker G, Boyer M, Gallagher M. Severe tinnitus and its effect on selective and divided attention. Int J Audiol. 2007 May;46(5):208-16. doi: 10.1080/14992020601102329. PMID 17487668
- [Background] Rossiter S, Stevens C, Walker G. Tinnitus and its effect on working memory and attention. J Speech Lang Hear Res. 2006 Feb;49(1):150-60. doi: 10.1044/1092-4388(2006/012). PMID 16533080
- [Background] Namas R, Ghuma A, Hermus L, Zamora R, Okonkwo DO, Billiar TR, Vodovotz Y. The acute inflammatory response in trauma / hemorrhage and traumatic brain injury: current state and emerging prospects. Libyan J Med. 2009 Sep 1;4(3):97-103. doi: 10.4176/090325. PMID 21483522
- [Background] Eyre H, Baune BT. Neuroplastic changes in depression: a role for the immune system. Psychoneuroendocrinology. 2012 Sep;37(9):1397-416. doi: 10.1016/j.psyneuen.2012.03.019. Epub 2012 Apr 21. PMID 22525700
- [Background] Beattie EC, Stellwagen D, Morishita W, Bresnahan JC, Ha BK, Von Zastrow M, Beattie MS, Malenka RC. Control of synaptic strength by glial TNFalpha. Science. 2002 Mar 22;295(5563):2282-5. doi: 10.1126/science.1067859. PMID 11910117
- [Background] Steinmetz CC, Turrigiano GG. Tumor necrosis factor-alpha signaling maintains the ability of cortical synapses to express synaptic scaling. J Neurosci. 2010 Nov 3;30(44):14685-90. doi: 10.1523/JNEUROSCI.2210-10.2010. PMID 21048125
- [Background] Stellwagen D, Malenka RC. Synaptic scaling mediated by glial TNF-alpha. Nature. 2006 Apr 20;440(7087):1054-9. doi: 10.1038/nature04671. Epub 2006 Mar 19. PMID 16547515
- [Background] Schaette R, Kempter R. Computational models of neurophysiological correlates of tinnitus. Front Syst Neurosci. 2012 May 8;6:34. doi: 10.3389/fnsys.2012.00034. eCollection 2012. PMID 22586377
- [Background] Yang S, Bao S. Homeostatic mechanisms and treatment of tinnitus. Restor Neurol Neurosci. 2013;31(2):99-108. doi: 10.3233/RNN-120248. PMID 23435453
- [Background] Yang S, Weiner BD, Zhang LS, Cho SJ, Bao S. Homeostatic plasticity drives tinnitus perception in an animal model. Proc Natl Acad Sci U S A. 2011 Sep 6;108(36):14974-9. doi: 10.1073/pnas.1107998108. Epub 2011 Sep 6. PMID 21896771
- [Background] Weinberg MS, Blake BL, McCown TJ. Opposing actions of hippocampus TNFalpha receptors on limbic seizure susceptibility. Exp Neurol. 2013 Sep;247:429-37. doi: 10.1016/j.expneurol.2013.01.011. Epub 2013 Jan 16. PMID 23333565
- [Background] Kaneko M, Stellwagen D, Malenka RC, Stryker MP. Tumor necrosis factor-alpha mediates one component of competitive, experience-dependent plasticity in developing visual cortex. Neuron. 2008 Jun 12;58(5):673-80. doi: 10.1016/j.neuron.2008.04.023. PMID 18549780
- [Background] Stellwagen D, Beattie EC, Seo JY, Malenka RC. Differential regulation of AMPA receptor and GABA receptor trafficking by tumor necrosis factor-alpha. J Neurosci. 2005 Mar 23;25(12):3219-28. doi: 10.1523/JNEUROSCI.4486-04.2005. PMID 15788779
- [Background] Ogoshi F, Yin HZ, Kuppumbatti Y, Song B, Amindari S, Weiss JH. Tumor necrosis-factor-alpha (TNF-alpha) induces rapid insertion of Ca2+-permeable alpha-amino-3-hydroxyl-5-methyl-4-isoxazole-propionate (AMPA)/kainate (Ca-A/K) channels in a subset of hippocampal pyramidal neurons. Exp Neurol. 2005 Jun;193(2):384-93. doi: 10.1016/j.expneurol.2004.12.026. PMID 15869941
- [Background] Llano DA, Turner J, Caspary DM. Diminished cortical inhibition in an aging mouse model of chronic tinnitus. J Neurosci. 2012 Nov 14;32(46):16141-8. doi: 10.1523/JNEUROSCI.2499-12.2012. PMID 23152598
- [Background] Middleton JW, Kiritani T, Pedersen C, Turner JG, Shepherd GM, Tzounopoulos T. Mice with behavioral evidence of tinnitus exhibit dorsal cochlear nucleus hyperactivity because of decreased GABAergic inhibition. Proc Natl Acad Sci U S A. 2011 May 3;108(18):7601-6. doi: 10.1073/pnas.1100223108. Epub 2011 Apr 18. PMID 21502491
- [Background] Brozoski T, Odintsov B, Bauer C. Gamma-aminobutyric acid and glutamic acid levels in the auditory pathway of rats with chronic tinnitus: a direct determination using high resolution point-resolved proton magnetic resonance spectroscopy (H-MRS). Front Syst Neurosci. 2012 Feb 24;6:9. doi: 10.3389/fnsys.2012.00009. eCollection 2012. PMID 22383901
- [Background] Isaacson JE, Moyer MT, Schuler HG, Blackall GF. Clinical associations between tinnitus and chronic pain. Otolaryngol Head Neck Surg. 2003 May;128(5):706-10. doi: 10.1016/S0194-59980300227-4. PMID 12748565
- [Background] Moller AR. Similarities between chronic pain and tinnitus. Am J Otol. 1997 Sep;18(5):577-85. PMID 9303153
- [Background] Tonndorf J. The analogy between tinnitus and pain: a suggestion for a physiological basis of chronic tinnitus. Hear Res. 1987;28(2-3):271-5. doi: 10.1016/0378-5955(87)90054-2. PMID 2820913
- [Background] De Ridder D, Elgoyhen AB, Romo R, Langguth B. Phantom percepts: tinnitus and pain as persisting aversive memory networks. Proc Natl Acad Sci U S A. 2011 May 17;108(20):8075-80. doi: 10.1073/pnas.1018466108. Epub 2011 Apr 18. PMID 21502503
- [Background] Ignatowski TA, Covey WC, Knight PR, Severin CM, Nickola TJ, Spengler RN. Brain-derived TNFalpha mediates neuropathic pain. Brain Res. 1999 Sep 11;841(1-2):70-7. doi: 10.1016/s0006-8993(99)01782-5. PMID 10546989
- [Background] Covey WC, Ignatowski TA, Knight PR, Spengler RN. Brain-derived TNFalpha: involvement in neuroplastic changes implicated in the conscious perception of persistent pain. Brain Res. 2000 Mar 17;859(1):113-22. doi: 10.1016/s0006-8993(00)01965-x. PMID 10720620
- [Background] Hess A, Axmann R, Rech J, Finzel S, Heindl C, Kreitz S, Sergeeva M, Saake M, Garcia M, Kollias G, Straub RH, Sporns O, Doerfler A, Brune K, Schett G. Blockade of TNF-alpha rapidly inhibits pain responses in the central nervous system. Proc Natl Acad Sci U S A. 2011 Mar 1;108(9):3731-6. doi: 10.1073/pnas.1011774108. Epub 2011 Jan 18. PMID 21245297
- [Background] Widomski D, Fretland DJ, Gasiecki AF, Collins PW. The prostaglandin analogs, misoprostol and SC-46275, potently inhibit cytokine release from activated human monocytes. Immunopharmacol Immunotoxicol. 1997 May;19(2):165-74. doi: 10.3109/08923979709007656. PMID 9130003
- [Background] Briner W, House J, O'Leary M. Synthetic prostaglandin E1 misoprostol as a treatment for tinnitus. Arch Otolaryngol Head Neck Surg. 1993 Jun;119(6):652-4. doi: 10.1001/archotol.1993.01880180068013. PMID 8499097
- [Background] Akkuzu B, Yilmaz I, Cakmak O, Ozluoglu LN. Efficacy of misoprostol in the treatment of tinnitus in patients with diabetes and/or hypertension. Auris Nasus Larynx. 2004 Sep;31(3):226-32. doi: 10.1016/j.anl.2004.03.005. PMID 15364356
- [Background] Page TH, Turner JJ, Brown AC, Timms EM, Inglis JJ, Brennan FM, Foxwell BM, Ray KP, Feldmann M. Nonsteroidal anti-inflammatory drugs increase TNF production in rheumatoid synovial membrane cultures and whole blood. J Immunol. 2010 Sep 15;185(6):3694-701. doi: 10.4049/jimmunol.1000906. Epub 2010 Aug 16. PMID 20713883
- [Background] Hwang JH, Chen JC, Yang SY, Wang MF, Chan YC. Expression of tumor necrosis factor-alpha and interleukin-1beta genes in the cochlea and inferior colliculus in salicylate-induced tinnitus. J Neuroinflammation. 2011 Apr 9;8:30. doi: 10.1186/1742-2094-8-30. PMID 21477330
- [Background] Wang HT, Luo B, Zhou KQ, Xu TL, Chen L. Sodium salicylate reduces inhibitory postsynaptic currents in neurons of rat auditory cortex. Hear Res. 2006 May;215(1-2):77-83. doi: 10.1016/j.heares.2006.03.004. Epub 2006 Apr 24. PMID 16632286
- [Background] Satoh H, Firestein GS, Billings PB, Harris JP, Keithley EM. Tumor necrosis factor-alpha, an initiator, and etanercept, an inhibitor of cochlear inflammation. Laryngoscope. 2002 Sep;112(9):1627-34. doi: 10.1097/00005537-200209000-00019. PMID 12352677
- [Background] Wang X, Truong T, Billings PB, Harris JP, Keithley EM. Blockage of immune-mediated inner ear damage by etanercept. Otol Neurotol. 2003 Jan;24(1):52-7. doi: 10.1097/00129492-200301000-00012. PMID 12544029
- [Background] Matteson EL, Choi HK, Poe DS, Wise C, Lowe VJ, McDonald TJ, Rahman MU. Etanercept therapy for immune-mediated cochleovestibular disorders: a multi-center, open-label, pilot study. Arthritis Rheum. 2005 Jun 15;53(3):337-42. doi: 10.1002/art.21179. PMID 15934127
- [Background] Rahman MU, Poe DS, Choi HK. Etanercept therapy for immune-mediated cochleovestibular disorders: preliminary results in a pilot study. Otol Neurotol. 2001 Sep;22(5):619-24. doi: 10.1097/00129492-200109000-00010. PMID 11568668
- [Background] Van Wijk F, Staecker H, Keithley E, Lefebvre PP. Local perfusion of the tumor necrosis factor alpha blocker infliximab to the inner ear improves autoimmune neurosensory hearing loss. Audiol Neurootol. 2006;11(6):357-65. doi: 10.1159/000095897. Epub 2006 Sep 21. PMID 16988499
- [Background] Scherer EQ, Yang J, Canis M, Reimann K, Ivanov K, Diehl CD, Backx PH, Wier WG, Strieth S, Wangemann P, Voigtlaender-Bolz J, Lidington D, Bolz SS. Tumor necrosis factor-alpha enhances microvascular tone and reduces blood flow in the cochlea via enhanced sphingosine-1-phosphate signaling. Stroke. 2010 Nov;41(11):2618-24. doi: 10.1161/STROKEAHA.110.593327. Epub 2010 Oct 7. PMID 20930159
- [Background] Hiller W, Goebel G. A psychometric study of complaints in chronic tinnitus. J Psychosom Res. 1992 May;36(4):337-48. doi: 10.1016/0022-3999(92)90070-i. PMID 1593509
- [Background] Falkenberg ES, Wie OB. Anxiety and depression in tinnitus patients: 5-year follow-up assessment after completion of habituation therapy. Int J Otolaryngol. 2012;2012:375460. doi: 10.1155/2012/375460. Epub 2012 Mar 28. PMID 22536254
- [Background] Halford JB, Anderson SD. Anxiety and depression in tinnitus sufferers. J Psychosom Res. 1991;35(4-5):383-90. doi: 10.1016/0022-3999(91)90033-k. PMID 1920169
- [Background] Harrop-Griffiths J, Katon W, Dobie R, Sakai C, Russo J. Chronic tinnitus: association with psychiatric diagnoses. J Psychosom Res. 1987;31(5):613-21. doi: 10.1016/0022-3999(87)90040-7. PMID 3430424
- [Background] Henry JL, Wilson PH. Coping with Tinnitus: Two Studies of Psychological and Audiological Characteristics of Patients with High and Low Tinnitus-Related Distress. Int Tinnitus J. 1995;1(2):85-92. PMID 10753328
- [Background] Seydel C, Haupt H, Olze H, Szczepek AJ, Mazurek B. Gender and chronic tinnitus: differences in tinnitus-related distress depend on age and duration of tinnitus. Ear Hear. 2013 Sep;34(5):661-72. doi: 10.1097/AUD.0b013e31828149f2. PMID 23439056
- [Background] Tyler RS, Gogel SA, Gehringer AK. Tinnitus activities treatment. Prog Brain Res. 2007;166:425-34. doi: 10.1016/S0079-6123(07)66041-5. PMID 17956807
- [Background] Tyler R, Ji H, Perreau A, Witt S, Noble W, Coelho C. Development and validation of the tinnitus primary function questionnaire. Am J Audiol. 2014 Sep;23(3):260-72. doi: 10.1044/2014_AJA-13-0014. PMID 24811293
- [Background] Scott B, Lindberg P, Melin L, Lyttkens L. Predictors of tinnitus discomfort, adaptation and subjective loudness. Br J Audiol. 1990 Feb;24(1):51-62. doi: 10.3109/03005369009077842. PMID 2317601
- [Background] Herbert TB, Cohen S. Stress and immunity in humans: a meta-analytic review. Psychosom Med. 1993 Jul-Aug;55(4):364-79. doi: 10.1097/00006842-199307000-00004. PMID 8416086
- [Background] Kiecolt-Glaser JK, Marucha PT, Malarkey WB, Mercado AM, Glaser R. Slowing of wound healing by psychological stress. Lancet. 1995 Nov 4;346(8984):1194-6. doi: 10.1016/s0140-6736(95)92899-5. PMID 7475659
- [Background] Huerta PT, Kowal C, DeGiorgio LA, Volpe BT, Diamond B. Immunity and behavior: antibodies alter emotion. Proc Natl Acad Sci U S A. 2006 Jan 17;103(3):678-83. doi: 10.1073/pnas.0510055103. Epub 2006 Jan 4. PMID 16407105
- [Background] Andrews JA, Neises KD. Cells, biomarkers, and post-traumatic stress disorder: evidence for peripheral involvement in a central disease. J Neurochem. 2012 Jan;120(1):26-36. doi: 10.1111/j.1471-4159.2011.07545.x. Epub 2011 Nov 17. PMID 22017326
- [Background] Hansel A, Hong S, Camara RJ, von Kanel R. Inflammation as a psychophysiological biomarker in chronic psychosocial stress. Neurosci Biobehav Rev. 2010 Sep;35(1):115-21. doi: 10.1016/j.neubiorev.2009.12.012. Epub 2009 Dec 22. PMID 20026349
- [Background] Steptoe A, Hamer M, Chida Y. The effects of acute psychological stress on circulating inflammatory factors in humans: a review and meta-analysis. Brain Behav Immun. 2007 Oct;21(7):901-12. doi: 10.1016/j.bbi.2007.03.011. Epub 2007 May 1. PMID 17475444
- [Background] Bob P, Raboch J, Maes M, Susta M, Pavlat J, Jasova D, Vevera J, Uhrova J, Benakova H, Zima T. Depression, traumatic stress and interleukin-6. J Affect Disord. 2010 Jan;120(1-3):231-4. doi: 10.1016/j.jad.2009.03.017. PMID 19359044
- [Background] Szczepek AJ, Haupt H, Klapp BF, Olze H, Mazurek B. Biological correlates of tinnitus-related distress: an exploratory study. Hear Res. 2014 Dec;318:23-30. doi: 10.1016/j.heares.2014.10.007. Epub 2014 Oct 28. PMID 25445818
- [Background] Weber C, Arck P, Mazurek B, Klapp BF. Impact of a relaxation training on psychometric and immunologic parameters in tinnitus sufferers. J Psychosom Res. 2002 Jan;52(1):29-33. doi: 10.1016/s0022-3999(01)00281-1. PMID 11801262
- [Background] Arck PC, Rose M, Hertwig K, Hagen E, Hildebrandt M, Klapp BF. Stress and immune mediators in miscarriage. Hum Reprod. 2001 Jul;16(7):1505-11. doi: 10.1093/humrep/16.7.1505. PMID 11425839
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Andersson G. Tinnitus loudness matchings in relation to annoyance and grading of severity. Auris Nasus Larynx. 2003 May;30(2):129-33. doi: 10.1016/s0385-8146(03)00008-7. PMID 12753982
- [Background] Andersson G, Lyttkens L, Larsen HC. Distinguishing levels of tinnitus distress. Clin Otolaryngol Allied Sci. 1999 Sep;24(5):404-10. doi: 10.1046/j.1365-2273.1999.00278.x. PMID 10542919

DOCUMENTS (1):
  • Informed Consent Form (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT04066348/ICF_003.pdf